CLINICAL TRIAL: NCT06862193
Title: The Effectiveneness of a Digital Intervention (the HM4MH-app) on Perinatal Psychological Wellbeing: Randomized Controlled Trial
Brief Title: Effectiveness of Digital Intervention (HM4MH-app) on Perinatal Psychological Wellbeing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristin Thomas, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM4MH
Record Dates: First submitted 2025-02-20; First posted 2025-03-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-10

CONDITIONS: Mobile Application; Behavior; Perinatal Mental Health
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HealthyMoms (control group) (Active Comparator): The control is a mobile application targeting women during the perinatal period, focusing on healthy lifestyles.
  Interventions: Behavioral: HealthyMoms
- Intervention: HealthyMoms4MentalHealth (Experimental): The intervention is a mobile application targeting women during the perinatal period, aiming to promote mental wellbeing.
  Interventions: Behavioral: HealthyMoms4MentalHealth

INTERVENTIONS:
Behavioral: HealthyMoms4MentalHealth — The intervention is a mobile application targeting women during the perinatal period, aiming to promote mental wellbeing.
  Arms: Intervention: HealthyMoms4MentalHealth
Behavioral: HealthyMoms — Digital intervention focusing on lifestyle behaviours during the perinatal period.
  Arms: HealthyMoms (control group)

SUMMARY:
As many as 25% of pregnant women report mental health problems such as depressiveness and anxiety. This is a major concern as mental illness during pregnancy can have severe and long-lasting consequences for the pregnant woman, the baby, as well as the partner. Digital interventions (e.g., apps) have shown to be promising in promoting mental wellbeing, at scale, however, the majority of tools have been developed and evaluated in a general population rather than tailored for pregnancy. The objective of this trial is to investigate the effectiveness of a new digital tool (HealthyMoms4MentalHealth-app) on mental health outcomes during the perinatal period.

DETAILED DESCRIPTION:
As many as 25% of pregnant women report mental health problems such as depressiveness and anxiety. This is a major concern as mental illness during pregnancy can have severe and long-lasting consequences for the pregnant woman, the baby, as well as the partner. Digital interventions (e.g., apps) have shown to be promising in promoting mental wellbeing, at scale, however, the majority of tools have been developed and evaluated in a general population rather than tailored for pregnancy. The objective of this trial is therefore to investigate the effectiveness of a new digital tool (HealthyMoms4MentalHealth-app) on mental health outcomes during the perinatal period. The tool has been developed tailored to the pregnancy and postpartum period.

The study is a two-arm parallel groups multi-centre randomised controlled trial where pregnant women (n=750) will be randomised (1:1) to either an intervention (HealthyMoms4MentalHealth-app) or control group (HealthyMoms-app). Primary outcome (mental wellbeing) and secondary outcomes (resilience, depressiveness, attachment, fear of childbirth) together with mediators (self-compassion and physical activity) will be measured at baseline (gestational week 10-12), timepoint 1 (gestational week 35-38) and timepoint 2 (8-10 weeks postpartum). Baseline will also assess demographic data (age, employment, education, birth country, living situation and number of children). Stressful life events will also be measured as potential confounding variable at baseline and timepoint 2 (8-10 weeks postpartum). In addition, information on obstetric and neonatal outcomes will be collected as continuous variables or incidence from medical records (Obstetrix®Cerner). They include gestational weight gain, caesarean section, infant birth weight and length and incidence of large-for gestational-age infant (birth weight >90th percentile for gestational age and gender).

ELIGIBILITY:
Inclusion Criteria:

(i) pregnant women attending a participating maternity health care centre who (ii) have access to their own mobile phone and BankID and is (iii) currently in gestational week 8-15 and (iv) is 18 years or older.

Exclusion Criteria:

* Previous psychotic disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Resilience | Baseline (gestational weeks 12-14); timepoint 1 (gestational week 35-37); timepoint 2 (8-9 weeks post-partum)
  Resilience will be measured using the Connor-Davidson Resilience Scale (CD-RISC-10) which includes 10 items graded on a five-point scale from "not at all true" to "almost always true". The items assess various aspects of resilience, such as emotional regulation, optimism, personal strength, and the ability to manage stress. Lower scores suggest lower resilience and possibly a greater vulnerability to stress and adversity whereas higher scores suggest higher resilience, meaning the individual is likely to be better equipped to handle stress or challenges.

SECONDARY OUTCOMES:
Depressive symptoms | Baseline (gestational week 12-14); timepoint 1 (gestational week 35-37); timepoint 2 (8-9 weeks post-partum)
  The Edinburgh Postpartum Depression Scale
  The Edinburgh Postpartum Depression Scale includes ten items graded on a four-point ordinal scale in which higher scores indicate increased depressive symptoms (range 0-30). The clinical cut-off used in Sweden for postpartum depression is >12.
Mental wellbeing | Baseline (gestational week 12-14); timepoint 1 (gestational week 35-37); timepoint 2 (8-9 weeks post-partum)
  Mental wellbeing will be measured with the Ryff Scales of Psychological Well-Being (RPWB), which includes 18 items. For this scale, higher scores indicate greater psychological well-being (range 18-108) and responses are given on a six-point Likert scale from "strongly disagree" to "strongly agree".
Prenatal attachment | Timepoint 1 (gestational week 35-37)
  Prenatal Attachment Inventory (PAI)
  Prenatal Attachment Inventory assess emotional attachment to the fetus using 21 items. Responses are made on a four-point likert scale and scores may range from 21 to 84 with higher scores indicating increased attachment quality/intensity.
Postpartum attachment | Timepoint 2 (8-9 weeks post-partum)
  Postpartum bonding questionnaire (PBQ)
  The Postpartum Bonding Questionnaire is a 25 item screening questionnaire for mother-infant bonding disorders. Items are rated on a 6-point scale ranging from "Always" to "Never."
Parental self-efficacy | Timepoint 2 (8-9 weeks post-partum)
  Parental self-efficacy
  The parental self-efficacy scale is a 17 item questionniare measuring parental self-efficacy with responses on a 7 point likert scale ranging from strongly disagree to strongly agree. Higher scores indicate higher self-reported parental self-efficacy.
Fear of childbirth | Mid-intervention (gestational week 32)
  Fear of childbirth (FOB)
  The the Fear of Birth Scale (FOBS) is a short instrument that measures fear of childbirth during pregnancy. It consists of two 100 mm Visual Analogue Scales (VAS) that are summed and averaged to get a score.

OTHER OUTCOMES:
Physical activity | Weekly registrations from enrollment until intervention completion (8-9 weeks post-partum).
  Physical activity, exercise, sedentary behaviour and screen time will be measured using six items. Two items are questions on the degree of physical activity during work and leisure time with a three-point response scale (sedentary to active). Four items are questions on the amount of time spent on screen time with a range from 0 to 14 hours weekly.
Self-compassion | Baseline (gestational week 12-14); timepoint 1 (gestational week 35-37); timepoint 2 (8-9 weeks post-partum) and mid-intervention (gestational week 18-19)
  The Self-Compassion Scale-Short Form (SCS-SF)
  The Self-Compassion Scale-Short Form (SCS-SF) is a 12-item scale graded on a five-point scale from "almost never" to "almost always". Self-compassion is measured in terms of self-kindness, self-judgment, common humanity, isolation, mindfulness and over identification.
Stressful life events | Baseline (gestational week 12-14); timepoint 2 (8-9 weeks post-partum)
  Stressful life events
  The Stressful Life Event Scale is a ten-item scale measuring life events such as divorce or health issues including when these events occurred (early life, during the last two years or never).

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Associate Professor Thomas, PhD, Principal Investigator — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Region Jönköping, Jönköping
  - Region Kalmar, Kalmar
  - Region Skåne, Malmo
  - Region Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided